CLINICAL TRIAL: NCT07117279
Title: A Prospective Observational Cohort Study on Dynamic CD8+ T-cell Profiling and Multi-omics Biomarkers for Predicting Conversion Therapy Response in Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhang Bi Xiang, MD, Professor, Tongji Hospital
Other Study IDs: TJ-IRB202506074
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to identify early predictors for successful liver cancer treatment conversion. We will track changes in immune cells (CD8+ T-cells) in the blood during chemotherapy infusion (HAIC/TACE) combined with targeted-immunotherapy for 120 patients with unresectable liver cancer. By analyzing blood and tissue samples at multiple timepoints using advanced cell profiling and multi-omics sequencing, we seek to:

Determine if early immune cell changes predict tumor shrinkage; Identify tissue biomarkers linked to longer recurrence-free survival; Build a personalized prediction model for treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-75 years) with histologically confirmed HCC
* At least one measurable lesion ≥10 mm
* Planned HAIC/TACE + immunotherapy regimen
* Child-Pugh class A liver function
* ECOG 0-1
* Signed informed consent

Exclusion Criteria:

* Prior systemic HCC therapy within 6 months
* Main portal vein tumor thrombosis (VP4)
* Active autoimmune disease requiring immunosuppression
* HIV/HBV/HCV with uncontrolled viral replication
* Pregnancy or refusal of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with unresectable liver cancer (HCC) who are scheduled to receive HAIC/TACE plus immunotherapy at major hospitals in Shanghai. All participants must have preserved liver function (Child-Pugh A) and at least one measurable tumor. Key requirements include willingness to undergo tumor biopsy before treatment and provide repeated blood samples during therapy. Expected recruitment sources: 1) Liver cancer specialty clinics (majority), 2) Interventional radiology units.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From treatment initiation to 12 weeks after first therapy cycle.
  Proportion of patients achieving tumor shrinkage (≥30% diameter reduction) or complete disappearance on CT/MRI scans, evaluated by RECIST v1.1 criteria. Complete response = 0 visible tumor; Partial response = ≥30% reduction in total tumor size.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | From surgery date to first recurrence or death (assessed monthly for 24 months).
  Time from successful tumor removal surgery to either: (a) new tumor growth on scans, or (b) death from any cause. Verified by quarterly CT/MRI + AFP testing.
Severe Treatment-Related Side Effects | From first treatment dose to 30 days after final dose.
  Number of patients experiencing grade ≥3 adverse events (e.g., liver damage, low blood counts) confirmed by lab tests and physician evaluation, using CTCAE v5.0 grading.